CLINICAL TRIAL: NCT00836355
Title: Pilot Study of Treatment With Intravenous Enoxaparin and/or Oral Minocycline to Limit Infarct Size After Ischemic Stroke
Brief Title: Enoxaparin and/or Minocycline in Acute Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too few acute stroke patients available to meet enrollment requirements.
Sponsor: NYU Langone Health (Other)
Collaborators: James N. Kirby Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-131
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-03

CONDITIONS: Acute Ischemic Stroke
Keywords: stroke; magnetic resonance imaging; enoxaparin; minocycline; NIH stroke scale; modified Rankin scale; neuroprotection
MeSH Terms: conditions — Ischemic Stroke; Stroke; cyclopia sequence | interventions — Enoxaparin; Minocycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Enoxaparin (Experimental)
  Interventions: Drug: Enoxaparin
- Minocycline (Experimental): Minocycline 200 mg orally once daily for 5 days
  Interventions: Drug: Minocycline
- Enoxaparin and minocycline (Experimental)
  Interventions: Drug: Enoxaparin; Drug: Minocycline
- Control (No Intervention)

INTERVENTIONS:
Drug: Enoxaparin — 2 (or 3) intravenous doses, the first on study entry, the last 24 hours later
  Other Names: Lovenox®
  Arms: Enoxaparin; Enoxaparin and minocycline
Drug: Minocycline — 200 mg orally once daily for 5 days
  Other Names: Minocin®
  Arms: Enoxaparin and minocycline; Minocycline

SUMMARY:
The purpose of this study is to investigate whether enoxaparin, minocycline, or both medications in combination may help in recovery from acute stroke.

Enoxaparin (brand name Lovenox®) is a medication approved for use in humans to prevent and to treat blood clots in deep veins in certain specific medical situations. Minocycline (brand name Minocin®) is a tetracycline antibiotic approved to treat a number of bacterial infections in humans. The investigators are studying these medications in acute human stroke because they have each been separately shown to reduce the amount of injured brain tissue in rats made to have acute ischemic stroke experimentally. In a human trial comparing minocycline with placebo (a sugar pill) acute ischemic stroke patients who took minocycline had better recovery after 1 week, 1 month and 3 months than patients who took placebo.

DETAILED DESCRIPTION:
Enoxaparin is a low molecular weight heparin (average molecular weight 4,500 daltons, vs. 12,000 to 15,000 daltons for unfractionated heparin) administered subcutaneously and intravenously. It is a marketed drug FDA-approved in various clinical situations for: the prevention and treatment of deep vein thrombosis; and in the treatment of acute myocardial infarction. Minocycline is an orally administered antibiotic of the tetracycline class. It is a marketed drug FDA-approved for the treatment of various bacterial and rickettsial infections. Both medications have been found to be neuroprotective in experimental stroke models. Minocycline has shown promise in a human acute stroke study.

This study is designed to investigate two logistically simple treatment regimens, singly or in combination, employing these medications for acute ischemic stroke:

1. pulsed intravenous (iv) administration of enoxaparin initiated within 6 hours and completed by 24 hours after stroke onset; and
2. oral minocycline treatment once daily for five days.

The goal of treatment is neuroprotection: the limitation of the loss of brain tissue that follows ischemic stroke.

ELIGIBILITY:
There are two Study Sections: A and B

--------------------------------------------

Study Section A Inclusion Criteria:

1. acute ischemic stroke in an adult in-patient who can complete screening and begin study treatment within 6 hours of stroke onset (onset time defined as the last time the patient was known to be at his/her usual level of functioning)
2. patient not a candidate for rTPA treatment because treatment cannot be started within the required 3 hours after stroke onset, or because rTPA treatment is refused.

Study Section A Exclusion Criteria:

1. intracranial hemorrhage;
2. subfalcine, transtentorial, or foramen magnum herniation on CT or MRI scan of the brain;
3. history of hypersensitivity or intolerance to or toxicity from enoxaparin, other heparinoids, heparin, minocycline, or other tetracyclines;
4. weight 125lbs or less;
5. active bleeding;
6. thrombolytic treatment or major surgery in the previous 24 hours;
7. anticipated need for treatment with coumarin, or a low-molecular weight heparin other than enoxaparin, or unfractionated heparin before 36 hours after stroke onset (but see deep venous thrombosis prophylaxis, below);
8. INR above the normal range;
9. known coagulopathy;
10. platelet count <100,000/mm3 (if the count drops below 100,000 while on enoxaparin, the medication will be stopped)
11. pregnancy or lactation;
12. undergoing dialysis; severe renal impairment (creatinine clearance known or estimated to be <30ml/min);
13. mean arterial BP (taken to be 1/3 of the difference in mm Hg between diastolic BP and systolic BP, added to the diastolic BP) of 130 mm Hg or greater; (if the mean arterial BP is 130 mm Hg or greater but can be reduced by treatment to < 130 mm Hg, with systolic BP in the 150 169 mm Hg range, the patient may be entered).

Patients in Study Section A will be randomly assigned to one of the four treatment arms: enoxaparin, minocycline, enoxaparin and minocycline, or no intervention.

--------------------------------------------

Study Section B Inclusion Criteria:

1. acute ischemic stroke in an adult in-patient who can complete screening and begin study treatment within 24 hours of stroke onset (onset time defined as the last time the patient was known to be at his/her usual level of functioning;)
2. patient does not qualify for, or declines to participate in, Study Section A.

Study Section B Exclusion Criteria:

1. acute primary intracranial hemorrhage;
2. subfalcine, transtentorial, or foramen magnum herniation on CT or MRI scan of the brain;
3. pregnancy or lactation.

Patients in Study Section B will be randomly assigned to one of TWO treatment arms: minocycline, or no intervention.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saran Jonas, M.D., Principal Investigator — Department of Neurology; New York University School of Medicine; Giacinto Grieco, M.D., Study Director — Department of Neurology; New York University School of Medicine
Locations (2):
- United States (2):
  - Bellevue Hospital Center, New York, New York
  - New York University Langone Medical Center, New York, New York

REFERENCES:
- [Background] Lampl Y, Boaz M, Gilad R, Lorberboym M, Dabby R, Rapoport A, Anca-Hershkowitz M, Sadeh M. Minocycline treatment in acute stroke: an open-label, evaluator-blinded study. Neurology. 2007 Oct 2;69(14):1404-10. doi: 10.1212/01.wnl.0000277487.04281.db. PMID 17909152
- [Background] Mary V, Wahl F, Uzan A, Stutzmann JM. Enoxaparin in experimental stroke: neuroprotection and therapeutic window of opportunity. Stroke. 2001 Apr;32(4):993-9. doi: 10.1161/01.str.32.4.993. PMID 11283402
- [Background] Quartermain D, Li Y, Jonas S. Enoxaparin, a low molecular weight heparin decreases infarct size and improves sensorimotor function in a rat model of focal cerebral ischemia. Neurosci Lett. 2000 Jul 14;288(2):155-8. doi: 10.1016/s0304-3940(00)01223-4. PMID 10876084
- [Background] Quartermain D, Li YS, Jonas S. The low molecular weight heparin enoxaparin reduces infarct size in a rat model of temporary focal ischemia. Cerebrovasc Dis. 2003;16(4):346-55. doi: 10.1159/000072556. PMID 13130175
- [Background] Xu L, Fagan SC, Waller JL, Edwards D, Borlongan CV, Zheng J, Hill WD, Feuerstein G, Hess DC. Low dose intravenous minocycline is neuroprotective after middle cerebral artery occlusion-reperfusion in rats. BMC Neurol. 2004 Apr 26;4:7. doi: 10.1186/1471-2377-4-7. PMID 15109399
- [Background] Yrjanheikki J, Tikka T, Keinanen R, Goldsteins G, Chan PH, Koistinaho J. A tetracycline derivative, minocycline, reduces inflammation and protects against focal cerebral ischemia with a wide therapeutic window. Proc Natl Acad Sci U S A. 1999 Nov 9;96(23):13496-500. doi: 10.1073/pnas.96.23.13496. PMID 10557349
- [Background] Liu Z, Fan Y, Won SJ, Neumann M, Hu D, Zhou L, Weinstein PR, Liu J. Chronic treatment with minocycline preserves adult new neurons and reduces functional impairment after focal cerebral ischemia. Stroke. 2007 Jan;38(1):146-52. doi: 10.1161/01.STR.0000251791.64910.cd. Epub 2006 Nov 22. PMID 17122429

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enoxaparin | Minocycline | Enoxaparin and Minocycline | Control
Started | 0 | 4 | 0 | 2
Completed | 0 | 4 | 0 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enoxaparin | Minocycline | Enoxaparin and Minocycline | Control | Total
Number analyzed (Participants) | 0 | 4 | 0 | 2 | 6
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 |  | 0 | 0
  Between 18 and 65 years |  | 4 |  | 1 | 5
  >=65 years |  | 0 |  | 1 | 1
Gender [Number; unit: participants]
  Female |  | 1 |  | 1 | 2
  Male |  | 3 |  | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Indices of Salvaged Ischemic Penumbra and of Final Infarct Volume Based on Quantitative Volumetric Analyses of Pre- and Post-treatment Perfusion-weighted and Diffusion-weighted Brain MR Imaging
Time Frame: Within approximately 7 days of stroke onset
Population: Although all participants completed the study, none of them had the necessary MRIs performed to gather outcome measure data. The study was closed once it was determined that logistically, it was not possible to complete the study at that point in time.
Arm/Group | Enoxaparin | Minocycline | Enoxaparin and Minocycline | Control
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: NIH Stroke Scale Scores
Time Frame: Baseline and after approximately one week
Population: This trial was terminated early because of logistical challenges in data collection. No outcome measures data was able to be collected.
Arm/Group | Enoxaparin | Minocycline | Enoxaparin and Minocycline | Control
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Modified Rankin Scale Score
Time Frame: Baseline, and approximately one week and 3 months later
Population: as for outcome 2
Arm/Group | Enoxaparin | Minocycline | Enoxaparin and Minocycline | Control
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Enoxaparin | Minocycline | Enoxaparin and Minocycline | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/4 | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/4 | 0/0 | 0/2

LIMITATIONS AND CAVEATS:
This trial was terminated early because of logistical challenges in data collection. No outcome measures data was able to be collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes